CLINICAL TRIAL: NCT02282007
Title: Norwegian Psychomotor Physiotherapy - The Effect on Quality of Life, The Feeling of Pain, Coping, Physical, Psychological and Social Functioning After the Treatment
Brief Title: Norwegian Psychomotor Physiotherapy - The Effect on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Astrid Bergland, Professor, Oslo Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REK 2013/1913
Record Dates: First submitted 2014-03-17; First posted 2014-11-04 (Estimated); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Pain; Stress; Psychosomatic Diseases; Muscle Skeletal Disorders
Keywords: Quality of life
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Intervention:Control group (No Intervention)
- Individual NPMP to the participants (Experimental): This arm will receive NPMP for 6 months, individually adjusted to their problems.
  Interventions: Behavioral: Individual NPMP to the participants

INTERVENTIONS:
Behavioral: Individual NPMP to the participants — The participants in the intervention group will receive NPMP individually adjusted for six months. NPMP is not a standardized treatment approach, but individually adjusted to the individual patient according to their individual problems.
  Arms: Individual NPMP to the participants

SUMMARY:
More and more people suffer from stress-related illness and ailments that can greatly affect the individual's experienced quality of life and sense of coping since pain, physical, mental and social functioning are closely linked. Many of these people will seek primary care for help, and thus be referred to the Norwegian psychomotor physiotherapy (NPMP) performed by physiotherapists in primary care.

Data shows that for the first three months of 2009, 42% of patients were referred to NPMP had a musculoskeletal diagnosis as the first diagnosis, often in the form of long-term and comprehensive pain problems. Many of the patients also had emotional difficulties, but without being diagnosed with mental illness. 23% of patients who were referred to NPMP had a psychiatric diagnosis as the first diagnosis. The full range of psychiatric diagnoses are represented, but the majority of patients were treated for anxiety and depression.

The investigators want to let people who have had NPMP treatment to consider what effect the treatment has given, measured by separate registrations of quality of life, pain, physical, mental and social functioning.

DETAILED DESCRIPTION:
The primary aim of this is project intends to evaluate the effect of Norwegian psychomotor physiotherapy (NPMP) on Health related Quality of Life measured by Short-form Health Survey (SF-36). The secondary aims are to evaluate the effect of Norwegian psychomotor physiotherapy (NPMP) on the variables Subjective Health Complaints Inventory (SHC); Hopkins 's Symptom Check List , Örebro Screening for musculo-skeletal pain ,Numeric Pain Rating Scale , Oslo Social Support Scale , Coping and The self-esteem scale"

The study design is based on the guidelines for randomized controlled trials presented in the CONSORT statement. The study will address to people who have had NPMP treatment approach, and they will be asked to consider what effect the treatment has given, measured by separate registrations of quality of life, pain, physical, mental and social functioning.

Participants Power calculation based on the primary outcome Short-form Health Survey (SF-36) proved that minimum 170 participants must be recruited. The participants will be recruited among patients on the waiting list for NPMP by all psychomotor physiotherapists who are members of the Norwegian Physiotherapists Association. If patients want to participate in the study, they will be randomized to an intervention group and a control group by drawing lots.

The intervention group will have NPMP as usual in 6 months. The control group remains on the waiting list for 6 months. Participants in both groups will be asked to fill out the self-assessment questionnaire at the start of the project and at the completion of the project after six months. Participants in the intervention group will receive the same form after 12 months, to examine whether there have been any subsequent change after completion NPMF.

Timing of surveys:

Participants will be given questionnaires by the NPMP physiotherapist at

* Baseline - 2 weeks before NPMF (both groups)
* After 6 months (both groups)
* After 12 months (intervention group).

ELIGIBILITY:
Inclusion Criteria:

1. Being referred to NPMP
2. Being able to give informed consent
3. The therapist finds the NPMP to be a proper treatment to this patient

Exclusion Criteria:

1. Do not understand Norwegian

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-02; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Short-form Health Survey (SF-36) at 6 months | 6 months
  This will be assessed for both the control group and the intervention group.
Change from baseline in Short-form Health Survey (SF-36) at 12 months | 12 months
  This outcome measure will be assessed only for the intervention group.

SECONDARY OUTCOMES:
Change from baseline in Subjective Health Complaints Inventory (SHC) at 6 months | 6 months
  This will be assessed for both the control group and the intervention group.
Change from baseline in Subjective Health Complaints Inventory (SHC) at 12 months | 12 months
  This outcome measure will be assessed only for the intervention group.
Change from baseline in Hopkins 's Symptom Check List (Lipman et al., 1979) at 6 months | 6 months
  This will be assessed for both the control group and the intervention group.
Change from baseline in Hopkins 's Symptom Check List (Lipman et al., 1979) at 12 months | 12 months
  This outcome measure will be assessed only for the intervention group.
Change from baseline in Örebro Screening for musculo-skeletal pain (Linton et al., 2011) at 6 months | 6 months
  This outcome measure will be assessed both for the Control Group and for the intervention group.
Change from baseline in Örebro Screening for musculo-skeletal pain (Linton et al., 2011) at 12 months | 12 months
  This outcome measure will be assessed only for the intervention group.

OTHER OUTCOMES:
Change from baseline in Numeric Pain Rating Scale (NPRS) at 6 months | 6 months
  This outcome measure will be assessed both for the Control Group and for the intervention group.
Change from baseline in Numeric Pain Rating Scale (NPRS) at 12 months | 12 months
  This outcome measure will be assessed only for the intervention group.
Change from Baseline in Oslo Social Support Scale (OSS-3) at 6 months | 6 months
  This outcome measure will be assessed both for the Control Group and for the intervention group.
Change from Baseline in Oslo Social Support Scale (OSS-3) at 12 months | 12 months
  This outcome measure will be assessed only for the intervention group.
Change from Baseline in Coping, (Pearlin & Schooler, 1978) at 6 months | 6 months
  This outcome measure will be assessed both for the Control Group and for the intervention group.
Change from Baseline in Coping, (Pearlin & Schooler, 1978) at 12 months | 12 months
  This outcome measure will be assessed only for the intervention group.
Change from Baseline in The self-esteem scale" (Rosenberg 1965) at 6 months | 6 months
  This outcome measure will be assessed both for the Control Group and for the intervention group.
Change from Baseline in The self-esteem scale" (Rosenberg 1965) at 12 months | 12 months
  This outcome measure will be assessed only for the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid Bergland, Phd, Principal Investigator — Oslo Metropolitan University
Locations (2):
- Norway (2):
  - Oslo and Akershus University College of Applied Sciences, Oslo
  - HIOA, Oslo